CLINICAL TRIAL: NCT03335800
Title: Apple Heart Study: Assessment of Wristwatch-Based Photoplethysmography to Identify Cardiac Arrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apple Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Minang (Mintu) Turakhia, Associate Professor of Medicine, Stanford University, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1.0
Record Dates: First submitted 2017-11-02; First posted 2017-11-08 (Actual); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Apple Heart Study App (Experimental)
  Interventions: Device: Apple Heart Study App

INTERVENTIONS:
Device: Apple Heart Study App — The Apple Heart Study app is a mobile medical app that analyzes pulse rate data. The app identifies episodes of irregular heart rhythms consistent with atrial fibrillation and other arrhythmias.

SUMMARY:
The Apple Heart Study (AHS) is a research study conducted to evaluate whether the Apple Heart Study App can use data collected on the Apple Watch to identify irregular heart rhythms, including those from potentially serious heart conditions such as atrial fibrillation. Up to 500,000 can participate in the study.

ELIGIBILITY:
Inclusion Criteria:

Possession of the following at time of eligibility screening, ascertained from automatic hardware/software/device pairing check:

* iPhone (5s or later) with iOS version 11.0 or later defined as iPhone model/iOS version used to complete screening eligibility.
* Apple Watch (Series 1 or later) with watchOS version 4.0 or later defined as Apple Watch model/watchOS paired with iPhone used to complete screening eligibility.
* Current resident of the United States at time of eligibility screening, defined by self-reported state of residence within the 50 states of the United States or District of Columbia.
* Proficient in written and spoken English, defined by self-report of comfort reading, writing, and speaking English on iPhone.
* Valid phone number associated with iPhone, ascertained from self-report.
* Valid email address, ascertained from self-report.

Exclusion Criteria:

* Self-reported diagnosis of Atrial Fibrillation.
* Self-reported diagnosis of Atrial Flutter.
* Currently on anti-coagulation therapy.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 419927 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minang (Mintu) Turakhia, MD, MAS, Principal Investigator — Stanford University; Marco V. Perez, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen KT, Yu J, Hedlin H, Phillips AT, Desai S, Cheung L, Kowey PR, Jain SS, Rumsfeld JS, Russo AM, Granger CB, Hills MT, Desai M, Mahaffey KW, Turakhia MP, Perez MV. Racial and Ethnic Representation and Study Engagement in a Siteless Digital Clinical Trial Using a Smartwatch: Findings From the Apple Heart Study. Mayo Clin Proc Digit Health. 2025 Jun 3;3(3):100232. doi: 10.1016/j.mcpdig.2025.100232. eCollection 2025 Sep. PMID 40673279
- [Derived] Garcia A, Balasubramanian V, Lee J, Gardner R, Gummidipundi S, Hung G, Ferris T, Cheung L, Granger C, Kowey P, Rumsfeld J, Russo A, Hills MT, Talati N, Nag D, Stein J, Tsay D, Desai S, Mahaffey K, Turakhia M, Perez M, Hedlin H, Desai M. Lessons learned in the Apple Heart Study and implications for the data management of future digital clinical trials. J Biopharm Stat. 2022 May 4;32(3):496-510. doi: 10.1080/10543406.2022.2080698. Epub 2022 Jun 12. PMID 35695137
- [Derived] Perez MV, Mahaffey KW, Hedlin H, Rumsfeld JS, Garcia A, Ferris T, Balasubramanian V, Russo AM, Rajmane A, Cheung L, Hung G, Lee J, Kowey P, Talati N, Nag D, Gummidipundi SE, Beatty A, Hills MT, Desai S, Granger CB, Desai M, Turakhia MP; Apple Heart Study Investigators. Large-Scale Assessment of a Smartwatch to Identify Atrial Fibrillation. N Engl J Med. 2019 Nov 14;381(20):1909-1917. doi: 10.1056/NEJMoa1901183. PMID 31722151
- [Derived] Turakhia MP, Desai M, Hedlin H, Rajmane A, Talati N, Ferris T, Desai S, Nag D, Patel M, Kowey P, Rumsfeld JS, Russo AM, Hills MT, Granger CB, Mahaffey KW, Perez MV. Rationale and design of a large-scale, app-based study to identify cardiac arrhythmias using a smartwatch: The Apple Heart Study. Am Heart J. 2019 Jan;207:66-75. doi: 10.1016/j.ahj.2018.09.002. Epub 2018 Sep 8. PMID 30392584
- See also: Website for study information — http://med.stanford.edu/appleheartstudy.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants downloaded the app; those with irregular pulse notification had a first teleconference visit with telehealth provider; an ECG patch was shipped to eligible participants to wear for 7 days, then they returned the patch for analysis and had a second teleconference visit to review the findings with the telehealth provider.
Groups:
- Apple Heart Study (AHS) App Users: Participants used the AHS App to detect episodes of irregular heart rhythms consistent with atrial fibrillation and other arrhythmias.
Period: Overall Study
Arm/Group | Apple Heart Study (AHS) App Users
Started | 419927
Received Irregular Pulse Notification | 2161
Attended First Study Visit | 945
ECG Patch Shipped | 658
ECG Patch Returned for Analysis | 450
Attended Second Study Visit | 396
Completed | 396
Not Completed | 419531

BASELINE CHARACTERISTICS:
Arm/Group | Apple Heart Study (AHS) App Users
Number analyzed (Participants) | 419927
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (13)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 177087
  Male | 238700
  Other | 396
  Not Reported | 3114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 286190
  Hispanic | 48775
  Black | 32275
  Asian | 26156
  American Indian | 4696
  Pacific Islander | 1493
  Middle Eastern | 3652
  Other or mixed race | 7958
  Not Reported | 8102
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 419927

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation (AF) of Greater Than 30 Seconds
Description: Proportion of notified participants who received an irregular pulse notification and that had AF detected on the ambulatory ECG.
Time Frame: During ambulatory ECG monitoring (up to 8 days)
Population: Participant who returned ECG Patch
Measure: Number (97.5% Confidence Interval); unit: Proportion of participants
Arm/Group | Apple Heart Study (AHS) App Users
Number analyzed (Participants) | 450
Proportion of participants | 0.34 [0.29 to 0.39]

2. Primary Outcome: Confirmed AF With a Detection by a Component of the App
Description: Simultaneous ambulatory ECG monitoring indicating an irregular rhythm consistent with AF during time intervals when an app component (tachogram) is positive for an irregular pulse among those who received an irregular heartbeat notification.
Time Frame: During ambulatory ECG monitoring (up to 8 days)
Measure: Number (97.5% Confidence Interval); unit: Proportion of Tachograms with AF
Units Other Than Participants: Tachograms
Arm/Group | Apple Heart Study (AHS) App Users
Number analyzed (Participants) | 450
Number analyzed (Tachograms) | 2089
Proportion of Tachograms with AF | 0.71 [0.69 to 0.74]

3. Secondary Outcome: Concordant AF With App Algorithm Notification
Description: Simultaneous ambulatory ECG monitoring indicating an irregular rhythm consistent with AF when the app based algorithm is positive for an irregular pulse among those who received a notification.
Time Frame: During ambulatory ECG monitoring (up to 8 days)
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Apple Heart Study (AHS) App Users
Number analyzed (Participants) | 86
Proportion of Participants | 0.84 [0.76 to 0.92]

4. Secondary Outcome: Self-reported Contact With a Health Care Provider
Description: Percentage of participant who self-reported contact with a health care provider within 90 days following an irregular pulse watch notification. Participants could self-report this health-care provider contact from 90 days following notification until the study survey went offline at end of study.
Time Frame: 90 days to 15 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Apple Heart Study (AHS) App Users
Number analyzed (Participants) | 1376
Percentage of participants | 57 [54 to 60]

ADVERSE EVENTS:
Time Frame: 1 year, 2 months and 14 days (participants may have reported adverse events at any time from enrollment to close of study)
Arm/Group | Apple Heart Study (AHS) App Users
All-Cause Mortality (participants affected / at risk) | 2/419927
Serious Adverse Events (participants affected / at risk) | 62/419927
Other Adverse Events (participants affected / at risk) | 0/419927
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apple Heart Study (AHS) App Users (N=419927)
Allergic reaction (Immune system disorders) | 1
Atrial Fibrilation (Cardiac disorders) | 40
Atrial Flutter (Cardiac disorders) | 1
Atrial Septal Defect diagnosed (Congenital, familial and genetic disorders) | 1
Chest Pain (Cardiac disorders) | 3
Chest Pain (General disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Death (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Drug Reaction (General disorders) | 1
Fall (General disorders) | 1
Increased frequency of Premature Ventricular Contractions (PVC) (Cardiac disorders) | 1
Left bundle branch block (Cardiac disorders) | 1
Mitral regurgitation (Cardiac disorders) | 1
Mitral Valve Disease (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Pneumonia (Infections and infestations) | 1
Procedural Complication (Surgical and medical procedures) | 1
Shortness of Breath (Cardiac disorders) | 1
Shortness of breath (Infections and infestations) | 1
Shortness of Breath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Stroke (Vascular disorders) | 1
Subdural hematoma (Vascular disorders) | 1
Syncope (Cardiac disorders) | 3
Trauma (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT03335800/Prot_SAP_000.pdf